CLINICAL TRIAL: NCT01693068
Title: A Multicenter, Open Label, Randomized Phase II Trial of the MEK Inhibitor Pimasertib or Dacarbazine in Previously Untreated Subjects With N-Ras Mutated Locally Advanced or Metastatic Malignant Cutaneous Melanoma
Brief Title: Phase II Trial of Pimasertib Versus Dacarbazine in N-Ras Mutated Cutaneous Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: EMD Serono (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMR 200066-007; 2012-002669-37 (EudraCT Number)
Record Dates: First submitted 2012-09-14; First posted 2012-09-26 (Estimated); Results first posted 2018-01-05 (Actual); Last update posted 2018-01-05 (Actual); Status verified 2017-12

CONDITIONS: N-Ras Mutated Locally Advanced or Metastasis Malignant Cutaneous Melanoma
Keywords: Cutaneous Melanoma; Dacarbazine; Pimasertib; N-Ras
MeSH Terms: conditions — Melanoma | interventions — N-(2,3-dihydroxypropyl)-1-((2-fluoro-4-iodophenyl)amino)isonicotinamide; Dacarbazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pimasertib (Experimental)
  Interventions: Drug: Pimasertib
- Dacarbazine (Active Comparator)
  Interventions: Drug: Dacarbazine

INTERVENTIONS:
Drug: Pimasertib — Subjects will receive pimasertib orally as monotherapy at a dose of 60 milligram (mg) twice daily continuously. Treatment will consist of repeated 21-day cycles which will continue until progression of the disease, unacceptable toxicity, withdrawal of informed consent, or death, whichever occurs first.
  Other Names: MSC1936369B; AS703026
  Arms: Pimasertib
Drug: Dacarbazine — Subjects will receive dacarbazine intravenously at dose of 1000 milligram per square meter (mg/m^2) of body surface area every 3 weeks on Day 1 of each 21-days cycle until progression of the disease, unacceptable toxicity, withdrawal of informed consent, or death, whichever occurs first. Eligible subjects with documented tumor progression on dacarbazine will offer to switch to pimasertib treatment.
  Arms: Dacarbazine

SUMMARY:
This is a Phase 2, multicenter, randomized, controlled, open-label trial of pimasertib versus dacarbazine aimed to confirm the activity of pimasertib in previously untreated subjects with N-Ras mutated locally advanced or metastatic malignant cutaneous melanoma by comparing the progression-free survival (PFS) of subjects treated with either pimasertib or dacarbazine and by getting a better understanding of the efficacy, safety, pharmacogenomics (PGx) and their relationship with pimasertib exposure.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with measurable, histologically or cytologically confirmed, locally advanced or metastatic cutaneous melanoma (stage III c or M1ac) N-Ras mutated. If N-Ras mutational status is unknown at screening, it must be prospectively defined before inclusion. If N-Ras mutational status is already known before screening, it must be retrospectively confirmed after inclusion by the sponsor.
* Tumor lesions amenable to biopsy or available tumor tissue as archival samples.
* Age greater than or equal to (>=) 18 years.
* Has read and understood the informed consent form and is willing and able to give informed consent. Fully understands requirements of the trial and willing to comply with all trial visits and assessments.
* Women of childbearing potential must have a negative blood pregnancy test at the screening visit. For the purposes of this trial, women of childbearing potential are defined as: "All female subjects after puberty unless they are post-menopausal for at least two years, or are surgically sterile".
* Female subjects of childbearing potential and male subjects with female partners of childbearing potential must be willing to avoid pregnancy by using an adequate method of contraception for 2 weeks prior to, during and four weeks after the last dose of trial medication. Effective contraception is defined as the method of contraception with a failure rate of less than 1% per year. Adequate contraception is defined as follows: two barrier methods or one barrier method with a spermicidal or intrauterine device or oral contraception for female partners of male subjects.

Exclusion Criteria:

* Has previous systemic treatment for locally advanced or metastatic cutaneous melanoma (excluding adjuvant treatment).
* Has non-measurable lesions, disease not evaluable by Response Evaluation Criteria in Solid Tumors (RECIST) v. 1.1
* Has an Eastern Cooperative Oncology Group performance status (ECOG PS) >1.
* Has bone marrow impairment as evidenced by Hemoglobin <10.0 g/dL, Neutrophil count <1.5 * 10^9/L, platelets <100 * 10^9/L.
* Has renal impairment as evidenced by calculated creatinine clearance <60 mL/min (according to the Cockcroft-Gault formula).
* Has liver function abnormality as defined by total bilirubin >1.5 * Upper Limit of Normal (ULN), or aspartate aminotransferase (AST)/alanine aminotransferase (ALT) >2.5 * ULN, for subjects with liver involvement AST/ALT >5 * ULN.
* Has significant cardiac conduction abnormalities, including QTc prolongation of >480 milliseconds and/or pacemaker or clinically relevant impaired cardiovascular function.
* Has hypertension uncontrolled by medication
* Has retinal degenerative disease (hereditary retinal degeneration or age-related macular degeneration), history of uveitis, or history of retinal vein occlusion (RVO) or any eye condition that would be considered a risk factor for RVO (e.g., uncontrolled glaucoma or ocular hypertension).
* Has known active central nervous system (CNS) metastases unless previously radiotherapy treated, stable by CT scan for at least 3 months without evidence of cerebral edema and no requirements for corticosteroids or anticonvulsants.
* History of difficulty swallowing, malabsorption or other chronic gastro-intestinal disease, or conditions that may hamper compliance and/or absorption of the tested product.
* Known human immunodeficiency virus (HIV) positivity, active hepatitis C, or active hepatitis B.
* Has undergone surgical intervention within 28 days from Day 1 of trial drug treatment.
* Has received extensive prior radiotherapy on more than 30% of bone marrow reserves, or prior bone marrow/stem cell transplantation within 5 years from Day 1 of trial drug treatment.
* Has history of any other significant medical disease such as major gastric or small bowel surgery, recent drainage of significant volumes of ascites or pleural effusion or has a psychiatric condition that might impair the subject well-being or preclude full participation in the trial.
* Has known hypersensitivity to dacarbazine.
* Is a pregnant or nursing female.
* Participated in another clinical trial within the past 28 days.
* Has creatine phosphokinase (CPK) level at baseline National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Grade >=2 (i.e > 2.5 * ULN), and/or has a previous history of myositis or rhabdomyolysis.
* Is suitable for treatment with an approved B-Raf inhibitor (exclusion criteria implemented in German amendment only).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2012-12-05 (Actual); Primary Completion 2015-07-04 (Actual); Study Completion 2016-10-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — EMD Serono Inc., a business of Merck KGaA, Darmstadt, Germany
Locations (101):
- United States (15):
  - Research Site, Birmingham, Alabama
  - Research Site, Tucson, Arizona
  - Research Site, San Francisco, California
  - Research Site, Miami Beach, Florida
  - Research Site, Orlando, Florida
  - Research Site, Maywood, Illinois
  - Research Site, Indianapolis, Indiana
  - Research Site, Boston, Massachusetts
  - Please contact the US Medical Information in, Rockland, Massachusetts
  - Research Site, St Louis, Missouri
  - Research Site, Morristown, New Jersey
  - Research Site, New York, New York
  - Research Site, Columbus, Ohio
  - Research Site, Dallas, Texas
  - Research Site, Madison, Wisconsin
- Australia (12):
  - Research Site, Adelaide, SA
  - Research Site, Albury/Wodonga
  - Research Site, Auchenflower
  - Research Site, Box Hill
  - Research Site, Greenslopes
  - Research Site, Herston
  - Research Site, Malvern
  - Research Site, North Sydney
  - Research Site, Prahran
  - Research Site, Wendouree
  - Research Site, Woodville South
  - Research site, Woolloongabba
- Belgium (2):
  - Research Site, Brussels
  - Research Site, Edegem
- France (13):
  - Research Site, Bordeaux
  - Research Site, Brest
  - Research Site, Dijon
  - Research Site, Lille
  - Research Site, Lyon
  - Research Site, Marseille
  - Research Site, Montpellier
  - Research Site, Nantes
  - Research Site, Paris
  - Research Site, Pierre-Bénite
  - Research Site, Rennes
  - Research Site, Toulouse
  - Research Site, Villejuif
- Germany (20):
  - Research Site, Augsburg
  - Research Site, Berlin
  - Research Site, Bonn
  - Research Site, Buxtehude
  - Research Site, Cologne
  - Research site, Düsseldorf
  - Research Site, Erlangen
  - Research Site, Essen
  - Research Site, Frankfurt am Main
  - Research Site, Hamburg
  - Research Site, Hanover
  - Research Site, Kiel
  - Research Site, Leipzig
  - Research Site, Magdeburg
  - Research Site, Mainz
  - Research site, München
  - Research Site, Münster
  - Research Site, Plauen
  - Research Site, Tübingen
  - Research Site, Würzburg
- Israel (3):
  - Research Site, Jerusalem
  - Research Site, Ramat Gan
  - Research Site, Tel Aviv
- Italy (8):
  - Research Site, Bari
  - Research Site, Genova
  - Research Site, Meldola - FC
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Padua
  - Research Site, Roma
  - Research Site, Siena
- Netherlands (3):
  - Research Site, Groningen
  - Research Site, Rotterdam
  - Research Site, Utrecht
- New Zealand (4):
  - Research Site, Christchurch
  - Research Site, Hamilton
  - Research Site, Palmerston North
  - Research Site, Tauranga
- South Africa (4):
  - Research Site, Durban
  - Research Site, Johannesburg
  - Research Site, Pietermaritzburg
  - Research Site, Pretoria
- Spain (8):
  - Research Site, Badalona
  - Research Site, Barcelona
  - Research Site, L'Hospitalet de Llobregat
  - Research Site, Madrid
  - Research Site, Majadahonda
  - Research Site, Málaga
  - Research Site, Pamplona
  - Research Site, Seville
- Sweden (2):
  - Research Site, Gothenburg
  - Research Site, Stockholm
- Switzerland (2):
  - Research Site, Basel
  - Research Site, Zurich
- United Kingdom (5):
  - Research Site, Cambridge
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Newcastle upon Tyne
  - Research Site, Southampton

REFERENCES:
- [Derived] Lebbe C, Dutriaux C, Lesimple T, Kruit W, Kerger J, Thomas L, Guillot B, Braud F, Garbe C, Grob JJ, Loquai C, Ferraresi V, Robert C, Vasey P, Conry R, Isaacs R, Espinosa E, Schueler A, Massimini G, Dreno B. Pimasertib Versus Dacarbazine in Patients With Unresectable NRAS-Mutated Cutaneous Melanoma: Phase II, Randomized, Controlled Trial with Crossover. Cancers (Basel). 2020 Jun 29;12(7):1727. doi: 10.3390/cancers12071727. PMID 32610581

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First/last subject (informed consent): 05 December 2012/04 June 2014. Cut-off date: 04 July 2015. Last subject last visit: 24 October 2016.
Pre-assignment Details: A total of 194 subjects were randomized in trial. Data presented based on the cut-off date of 04 July 2015.
Groups:
- Dacarbazine: Subjects received dacarbazine intravenously at dose of 1000 mg/m^2 of body surface area every 3 weeks on Day 1 of each 21-days cycle until progression of the disease, unacceptable toxicity, withdrawal of informed consent, or death, whichever occurred first. Eligible subjects with documented tumor progression on dacarbazine were offered to switch to pimasertib treatment.
- Pimasertib: Subjects received pimasertib orally as monotherapy at a dose of 60 milligram (mg) twice daily continuously. Treatment consisted of repeated 21-day cycles which was continued until progression of the disease, unacceptable toxicity, withdrawal of informed consent, or death, whichever occurred first.
- Pimasertib (Crossover): Subjects who were randomized and received dacarbazine and were allowed to crossover to pimasertib treatment on progression of their disease.
Period: Randomization Period
Arm/Group | Dacarbazine | Pimasertib | Pimasertib (Crossover)
Started | 64 | 130 | 0
Treated | 61 | 130 | 0
Completed | 62 | 125 | 0
Not Completed | 2 | 5 | 0
Not completed — On-study | 2 | 5 | 0
Period: Cross-over (Dacarbazine To Pimasertib)
Arm/Group | Dacarbazine | Pimasertib | Pimasertib (Crossover)
Started | 0 | 0 | 41
Treated | 0 | 0 | 41
Completed | 0 | 0 | 40
Not Completed | 0 | 0 | 1
Not completed — On-study | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) analysis set included all subjects who were randomized to trial treatment.
Groups:
- Pimasertib: Subjects received pimasertib orally as monotherapy at a dose of 60 mg twice daily continuously. Treatment consisted of repeated 21-day cycles which was continued until progression of the disease, unacceptable toxicity, withdrawal of informed consent, or death, whichever occurred first.
- Total: Total of all reporting groups
Arm/Group | Dacarbazine | Pimasertib | Total
Number analyzed (Participants) | 64 | 130 | 194
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 36 | 65 | 101
  >=65 years | 28 | 65 | 93
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 62 | 90
  Male | 36 | 68 | 104

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the duration (in weeks) from randomization until the first progressive disease (PD) observation as assessed by the Investigator according to Response Evaluation Criteria for Solid Tumors (RECIST) version 1.1, or death due to any cause when death occurred within 12 weeks after the last tumor assessment (otherwise censored), whichever occurred first. PD was defined as at least a 20% increase in the sum of diameters of the target lesions, taking as reference the smallest sum since the treatment started (including baseline), or appearance of one or more new lesions, and/or unequivocal progression of existing non-target lesions.
Time Frame: From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to cut-off date (04-Jul-2015)
Population: ITT analysis set included all subjects who were randomized to trial treatment.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Dacarbazine | Pimasertib
Number analyzed (Participants) | 64 | 130
weeks | 6.86 [6.00 to 12.14] | 13.00 [12.29 to 17.71]
Statistical Analysis 1: Comparison: Dacarbazine vs Pimasertib; Test type: Other — A log-rank test stratified by baseline Eastern Cooperative Oncology Group performance status (ECOG PS) (using the interactive voice response system [IVRS] value) will tested the null hypothesis of no difference between the Pimasertib (first line) and the Dacarbazine treatment groups at the 5% level; p = 0.0022, Stratified Log Rank Test; Hazard Ratio (HR) = 0.59, 95% CI 2-sided [0.42 to 0.83] — The Hazard Ratio is obtained from the Cox Proportional Hazards model based on dacarbazine and pimasertib only stratified by baseline ECOG Performance Status

2. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of subjects with complete response (CR) or partial response (PR) according to RECIST version 1.1 criteria. CR: defined as disappearance of all target and all non-target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to less than (<) 10 millimeter (mm). PR: defined as at least a 30% decrease in sum of diameters of target lesions, taking as reference the baseline sum diameters along with absence of new lesions and disease progression in non-target lesions.
Time Frame: as for outcome 1
Population: ITT analysis set included all subjects who were randomized to trial treatment.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Dacarbazine | Pimasertib
Number analyzed (Participants) | 64 | 130
percentage of subjects | 14.1 [6.6 to 25.0] | 26.9 [19.5 to 35.4]

3. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR was defined as the percentage of subjects with CR, PR, or stable disease (SD) for greater than (>) 3 months assessed by investigator according to RECIST version 1.1. CR: defined as disappearance of all target and all non-target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to less than <10 mm. PR: defined as at least a 30% decrease in sum of diameters of target lesions, taking as reference the baseline sum diameters along with absence of new lesions and disease progression in non-target lesions. SD: defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: as for outcome 1
Population: ITT analysis set included all subjects who were randomized to trial treatment.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Dacarbazine | Pimasertib
Number analyzed (Participants) | 64 | 130
percentage of subjects | 15.6 [7.8 to 26.9] | 33.1 [25.1 to 41.9]

4. Secondary Outcome: Percentage of Subjects With Progression-free Survival (PFS) at 6 Months
Description: PFS was defined as the duration (in weeks) from randomization until the first progressive disease (PD) observation as assessed by the Investigator according to Response Evaluation Criteria for Solid Tumors (RECIST) version 1.1, or death due to any cause when death occurred within 12 weeks after the last tumor assessment, whichever occurred first. PD was defined as at least a 20% increase in the sum of diameters of the target lesions, taking as reference the smallest sum since the treatment started (including baseline), or appearance of one or more new lesions, and/or unequivocal progression of existing non-target lesions. Percentage of Subjects with PFS at 6 Months were reported.
Time Frame: 6 months
Population: ITT analysis set included all subjects who were randomized to trial treatment.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Dacarbazine | Pimasertib
Number analyzed (Participants) | 64 | 130
percentage of subjects | 9.4 [3.6 to 18.6] | 17.3 [10.2 to 26.0]

5. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time (in months) from randomization to death due to any cause. Subjects without a death date were to be censored at the minimum of last known date alive, defined as the latest date available on the electronic case report form, and cut-off date.
Time Frame: From date of randomization until date of death from any cause, assessed up to cut-off date (04-Jul-2015)
Population: ITT analysis set included all subjects who were randomized to trial treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dacarbazine | Pimasertib
Number analyzed (Participants) | 64 | 130
months | 10.61 [7.26 to 16.49] | 8.87 [7.46 to 15.51]

6. Secondary Outcome: Percentage of Subjects With Overall Survival (OS) at 12 Months
Description: OS was defined as the time (in months) from randomization to death due to any cause. Subjects without a death date were to be censored at the minimum of last known date alive, defined as the latest date available on the electronic case report form, and cut-off date. Percentage of Subjects with OS at 12 months were reported.
Time Frame: 12 months
Population: ITT analysis set included all subjects who were randomized to trial treatment.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Dacarbazine | Pimasertib
Number analyzed (Participants) | 64 | 130
percentage of subjects | 44.5 [31.6 to 56.6] | 43.3 [34.5 to 51.8]

7. Secondary Outcome: Change From Baseline in Subject-reported Quality of Life Assessed by Functional Assessment Cancer Therapy - Melanoma Total Score (FACT-M TS) at Day 1 of Pre-Specified Cycles and End of Treatment (EOT)
Description: QoL assessed using Function Assessment Cancer Therapy-melanoma (FACT-M) assessment tool. This includes 27-item FACT-General (FACT-G) questionnaire which consists of 24 questions;7 relating to physical well-being (PWB),7 relating to social/family well-being (SWB),6 relating to emotional well-being (EWB) and 7 relating to functional well-being (FWB). Also, it includes melanoma-specific subscale consists of 16 questions for Melanoma Subscale (MS) and 8 questions for Melanoma Surgery Scale (MSS).Each of these questions could have a response of Not at all, a little bit, somewhat, quite a bit and very much. The responses were given a value between 0 and 4 with 4 being best response. The FACT-M Total Score (FACT-M TS) ranges from 0 to 172 and is derived as follows: FACT-M TS= PWB Score + SWB Score + EWB Score + FWB Score + MS Score. Higher scores represent a better quality of life.
Time Frame: Baseline, Day 1 of Cycle 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 19, 20, 21, 22, 23, 24, 25, 26, 27, 28, 30, 31, 32, 33, 35, 36, 37 and EOT (up to cut-off date [04-Jul-2015])
Population: ITT analysis set. Here "Number of Subjects Analyzed" = subjects evaluable for this outcome and "Number Analyzed" = subjects evaluable at specified time points for each arm, respectively. There were no subjects analyzed at certain time points (that is, Number Analyzed = 0) because there was no data collected for respective arms at those time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dacarbazine | Pimasertib
Number analyzed (Participants) | 58 | 126
units on a scale
  Baseline | 126.20 (23.828) | 132.24 (22.179)
  Change at Day 1 Cycle 2: number analyzed (Participants) | 45 | 99
  Change at Day 1 Cycle 2 | -3.05 (14.815) | -3.06 (18.492)
  Change at Day 1 Cycle 3: number analyzed (Participants) | 24 | 73
  Change at Day 1 Cycle 3 | 0.60 (19.965) | -6.77 (21.716)
  Change at Day 1 Cycle 4: number analyzed (Participants) | 23 | 63
  Change at Day 1 Cycle 4 | 4.11 (14.746) | -6.54 (19.919)
  Change at Day 1 Cycle 5: number analyzed (Participants) | 10 | 45
  Change at Day 1 Cycle 5 | 0.62 (11.810) | -2.81 (17.202)
  Change at Day 1 Cycle 6: number analyzed (Participants) | 9 | 33
  Change at Day 1 Cycle 6 | -3.71 (15.674) | -8.45 (20.939)
  Change at Day 1 Cycle 7: number analyzed (Participants) | 9 | 29
  Change at Day 1 Cycle 7 | -1.10 (13.318) | -8.84 (19.128)
  Change at Day 1 Cycle 8: number analyzed (Participants) | 8 | 18
  Change at Day 1 Cycle 8 | 1.28 (12.928) | -14.67 (18.508)
  Change at Day 1 Cycle 9: number analyzed (Participants) | 6 | 12
  Change at Day 1 Cycle 9 | 2.21 (16.224) | -13.67 (21.388)
  Change at Day 1 Cycle 10: number analyzed (Participants) | 6 | 10
  Change at Day 1 Cycle 10 | 4.40 (14.818) | -13.26 (20.716)
  Change at Day 1 Cycle 11: number analyzed (Participants) | 4 | 11
  Change at Day 1 Cycle 11 | 1.02 (19.161) | -14.10 (21.157)
  Change at Day 1 Cycle 12: number analyzed (Participants) | 4 | 11
  Change at Day 1 Cycle 12 | 1.56 (19.932) | -10.52 (18.895)
  Change at Day 1 Cycle 13: number analyzed (Participants) | 4 | 6
  Change at Day 1 Cycle 13 | 5.51 (20.191) | -13.38 (23.690)
  Change at Day 1 Cycle 14: number analyzed (Participants) | 2 | 8
  Change at Day 1 Cycle 14 | 11.50 (21.920) | -18.24 (22.998)
  Change at Day 1 Cycle 15: number analyzed (Participants) | 3 | 7
  Change at Day 1 Cycle 15 | 9.60 (15.345) | -11.33 (19.787)
  Change at Day 1 Cycle 16: number analyzed (Participants) | 3 | 7
  Change at Day 1 Cycle 16 | 10.56 (14.935) | -11.18 (23.680)
  Change at Day 1 Cycle 17: number analyzed (Participants) | 2 | 6
  Change at Day 1 Cycle 17 | 3.00 (5.657) | -9.18 (24.166)
  Change at Day 1 Cycle 18: number analyzed (Participants) | 1 | 5
  Change at Day 1 Cycle 18 | 27.00 (NA) — Standard deviation could not be estimated as there was only 1 subject analyzed at the specified time point. | -3.92 (9.640)
  Change at Day 1 Cycle 19: number analyzed (Participants) | 2 | 4
  Change at Day 1 Cycle 19 | 16.50 (14.849) | -1.15 (8.147)
  Change at Day 1 Cycle 20: number analyzed (Participants) | 2 | 3
  Change at Day 1 Cycle 20 | 16.00 (15.556) | 1.17 (5.947)
  Change at Day 1 Cycle 21: number analyzed (Participants) | 2 | 3
  Change at Day 1 Cycle 21 | 17.00 (14.142) | 4.17 (8.918)
  Change at Day 1 Cycle 22: number analyzed (Participants) | 2 | 3
  Change at Day 1 Cycle 22 | 18.00 (12.728) | 1.32 (11.163)
  Change at Day 1 Cycle 23: number analyzed (Participants) | 1 | 2
  Change at Day 1 Cycle 23 | 27.00 (NA) — Standard deviation could not be estimated as there was only 1 subject analyzed at the specified time point. | -13.69 (15.354)
  Change at Day 1 Cycle 24: number analyzed (Participants) | 2 | 1
  Change at Day 1 Cycle 24 | 13.50 (19.092) | -3.83 (NA) — Standard deviation could not be estimated as there was only 1 subject analyzed at the specified time point.
  Change at Day 1 Cycle 25: number analyzed (Participants) | 2 | 1
  Change at Day 1 Cycle 25 | 14.50 (17.678) | -3.83 (NA) — Standard deviation could not be estimated as there was only 1 subject analyzed at the specified time point.
  Change at Day 1 Cycle 26: number analyzed (Participants) | 1 | 1
  Change at Day 1 Cycle 26 | 27.00 (NA) — Standard deviation could not be estimated as there was only 1 subject analyzed at the specified time point. | -2.83 (NA) — Standard deviation could not be estimated as there was only 1 subject analyzed at the specified time point.
  Change at Day 1 Cycle 27: number analyzed (Participants) | 1 | 0
  Change at Day 1 Cycle 27 | 27.00 (NA) — Standard deviation could not be estimated as there was only 1 subject analyzed at the specified time point. |
  Change at Day 1 Cycle 28: number analyzed (Participants) | 1 | 1
  Change at Day 1 Cycle 28 | 27.00 (NA) — Standard deviation could not be estimated as there was only 1 subject analyzed at the specified time point. | -0.83 (NA) — Standard deviation could not be estimated as there was only 1 subject analyzed at the specified time point.
  Change at Day 1 Cycle 30: number analyzed (Participants) | 0 | 1
  Change at Day 1 Cycle 30 |  | -1.83 (NA) — Standard deviation could not be estimated as there was only 1 subject analyzed at the specified time point.
  Change at Day 1 Cycle 31: number analyzed (Participants) | 0 | 1
  Change at Day 1 Cycle 31 |  | -7.83 (NA) — Standard deviation could not be estimated as there was only 1 subject analyzed at the specified time point.
  Change at Day 1 Cycle 32: number analyzed (Participants) | 0 | 1
  Change at Day 1 Cycle 32 |  | -7.83 (NA) — Standard deviation could not be estimated as there was only 1 subject analyzed at the specified time point.
  Change at Day 1 Cycle 33: number analyzed (Participants) | 0 | 1
  Change at Day 1 Cycle 33 |  | -8.83 (NA) — Standard deviation could not be estimated as there was only 1 subject analyzed at the specified time point.
  Change at Day 1 Cycle 35: number analyzed (Participants) | 0 | 1
  Change at Day 1 Cycle 35 |  | -1.83 (NA) — Standard deviation could not be estimated as there was only 1 subject analyzed at the specified time point.
  Change at Day 1 Cycle 36: number analyzed (Participants) | 0 | 1
  Change at Day 1 Cycle 36 |  | -3.83 (NA) — Standard deviation could not be estimated as there was only 1 subject analyzed at the specified time point.
  Change at Day 1 Cycle 37: number analyzed (Participants) | 0 | 1
  Change at Day 1 Cycle 37 |  | -4.83 (NA) — Standard deviation could not be estimated as there was only 1 subject analyzed at the specified time point.
  Change at EOT: number analyzed (Participants) | 28 | 75
  Change at EOT | -7.91 (23.119) | -9.98 (20.560)

8. Secondary Outcome: Change From Baseline in Subject-reported Quality of Life Assessed by Functional Assessment Cancer Therapy - Melanoma Trial Outcome Index (FACT-M TOI) at Day 1 of Pre-Specified Cycles and End of Treatment (EOT)
Description: QoL assessed using FACT-M assessment tool. This includes 27-item FACT-G questionnaire which consists of 24 questions; 7 relating to PWB, 7 relating to SWB, 6 relating to EWB and 7 relating to FWB. Also, it includes melanoma-specific subscale consists of 16 questions for MS and 8 questions for the MSS. Each of these questions could have a response of Not at all, a little bit, somewhat, quite a bit and very much. The responses were given a value between 0 and 4 with 4 being best response. The FACT-M Trial Outcome Index (FACT-M TOI) ranges from 0 to a high of 120 and is derived as: FACT-M TOI = PWB Score + FWB Score +MS Score. Higher scores represent a better quality of life.
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dacarbazine | Pimasertib
Number analyzed (Participants) | 58 | 126
units on a scale
  Baseline | 90.35 (19.348) | 94.07 (17.534)
  Change at Day 1 Cycle 2: number analyzed (Participants) | 45 | 99
  Change at Day 1 Cycle 2 | -3.33 (12.015) | -4.40 (14.286)
  Change at Day 1 Cycle 3: number analyzed (Participants) | 24 | 73
  Change at Day 1 Cycle 3 | -0.69 (15.974) | -7.99 (17.089)
  Change at Day 1 Cycle 4: number analyzed (Participants) | 23 | 63
  Change at Day 1 Cycle 4 | 1.54 (10.304) | -7.97 (16.741)
  Change at Day 1 Cycle 5: number analyzed (Participants) | 10 | 45
  Change at Day 1 Cycle 5 | -0.86 (5.405) | -4.37 (14.084)
  Change at Day 1 Cycle 6: number analyzed (Participants) | 9 | 33
  Change at Day 1 Cycle 6 | -3.29 (7.752) | -9.15 (18.813)
  Change at Day 1 Cycle 7: number analyzed (Participants) | 9 | 29
  Change at Day 1 Cycle 7 | -2.07 (6.859) | -8.99 (14.783)
  Change at Day 1 Cycle 8: number analyzed (Participants) | 8 | 18
  Change at Day 1 Cycle 8 | 0.83 (5.161) | -15.09 (14.458)
  Change at Day 1 Cycle 9: number analyzed (Participants) | 6 | 12
  Change at Day 1 Cycle 9 | -1.93 (6.300) | -13.79 (17.198)
  Change at Day 1 Cycle 10: number analyzed (Participants) | 6 | 10
  Change at Day 1 Cycle 10 | -1.10 (5.654) | -12.37 (17.058)
  Change at Day 1 Cycle 11: number analyzed (Participants) | 4 | 11
  Change at Day 1 Cycle 11 | -2.90 (7.722) | -13.95 (17.006)
  Change at Day 1 Cycle 12: number analyzed (Participants) | 4 | 11
  Change at Day 1 Cycle 12 | -2.40 (7.408) | -11.95 (17.311)
  Change at Day 1 Cycle 13: number analyzed (Participants) | 4 | 6
  Change at Day 1 Cycle 13 | 0.80 (7.697) | -13.57 (21.699)
  Change at Day 1 Cycle 14: number analyzed (Participants) | 2 | 8
  Change at Day 1 Cycle 14 | 0.00 (4.243) | -18.55 (19.880)
  Change at Day 1 Cycle 15: number analyzed (Participants) | 3 | 7
  Change at Day 1 Cycle 15 | 1.60 (4.084) | -13.59 (15.747)
  Change at Day 1 Cycle 16: number analyzed (Participants) | 3 | 7
  Change at Day 1 Cycle 16 | 0.61 (3.994) | -13.15 (19.130)
  Change at Day 1 Cycle 17: number analyzed (Participants) | 2 | 6
  Change at Day 1 Cycle 17 | 2.50 (0.707) | -10.66 (20.007)
  Change at Day 1 Cycle 18: number analyzed (Participants) | 1 | 5
  Change at Day 1 Cycle 18 | 3.00 (NA) — Standard deviation could not be estimated as there was only 1 subject analyzed at the specified time point. | -5.72 (4.614)
  Change at Day 1 Cycle 19: number analyzed (Participants) | 2 | 4
  Change at Day 1 Cycle 19 | 2.50 (0.707) | -4.94 (5.238)
  Change at Day 1 Cycle 20: number analyzed (Participants) | 2 | 3
  Change at Day 1 Cycle 20 | 4.00 (1.414) | -2.33 (1.155)
  Change at Day 1 Cycle 21: number analyzed (Participants) | 2 | 3
  Change at Day 1 Cycle 21 | 3.50 (0.707) | 0.00 (2.000)
  Change at Day 1 Cycle 22: number analyzed (Participants) | 2 | 3
  Change at Day 1 Cycle 22 | 4.00 (1.414) | -1.40 (3.831)
  Change at Day 1 Cycle 23: number analyzed (Participants) | 1 | 2
  Change at Day 1 Cycle 23 | 3.00 (NA) — Standard deviation could not be estimated as there was only 1 subject analyzed at the specified time point. | -13.36 (16.061)
  Change at Day 1 Cycle 24: number analyzed (Participants) | 2 | 1
  Change at Day 1 Cycle 24 | 2.50 (0.707) | -2.00 (NA) — Standard deviation could not be estimated as there was only 1 subject analyzed at the specified time point.
  Change at Day 1 Cycle 25: number analyzed (Participants) | 2 | 1
  Change at Day 1 Cycle 25 | 3.50 (0.707) | -1.00 (NA) — Standard deviation could not be estimated as there was only 1 subject analyzed at the specified time point.
  Change at Day 1 Cycle 26: number analyzed (Participants) | 1 | 1
  Change at Day 1 Cycle 26 | 3.00 (NA) — Standard deviation could not be estimated as there was only 1 subject analyzed at the specified time point. | 0.00 (NA) — Standard deviation could not be estimated as there was only 1 subject analyzed at the specified time point.
  Change at Day 1 Cycle 27: number analyzed (Participants) | 1 | 0
  Change at Day 1 Cycle 27 | 3.00 (NA) — Standard deviation could not be estimated as there was only 1 subject analyzed at the specified time point. |
  Change at Day 1 Cycle 28: number analyzed (Participants) | 1 | 1
  Change at Day 1 Cycle 28 | 3.00 (NA) — Standard deviation could not be estimated as there was only 1 subject analyzed at the specified time point. | 1.00 (NA) — Standard deviation could not be estimated as there was only 1 subject analyzed at the specified time point.
  Change at Day 1 Cycle 30: number analyzed (Participants) | 0 | 1
  Change at Day 1 Cycle 30 |  | 1.00 (NA) — Standard deviation could not be estimated as there was only 1 subject analyzed at the specified time point.
  Change at Day 1 Cycle 31: number analyzed (Participants) | 0 | 1
  Change at Day 1 Cycle 31 |  | -3.00 (NA) — Standard deviation could not be estimated as there was only 1 subject analyzed at the specified time point.
  Change at Day 1 Cycle 32: number analyzed (Participants) | 0 | 1
  Change at Day 1 Cycle 32 |  | -4.00 (NA) — Standard deviation could not be estimated as there was only 1 subject analyzed at the specified time point.
  Change at Day 1 Cycle 33: number analyzed (Participants) | 0 | 1
  Change at Day 1 Cycle 33 |  | -3.00 (NA) — Standard deviation could not be estimated as there was only 1 subject analyzed at the specified time point.
  Change at Day 1 Cycle 35: number analyzed (Participants) | 0 | 1
  Change at Day 1 Cycle 35 |  | 0.00 (NA) — Standard deviation could not be estimated as there was only 1 subject analyzed at the specified time point.
  Change at Day 1 Cycle 36: number analyzed (Participants) | 0 | 1
  Change at Day 1 Cycle 36 |  | 0.00 (NA) — Standard deviation could not be estimated as there was only 1 subject analyzed at the specified time point.
  Change at Day 1 Cycle 37: number analyzed (Participants) | 0 | 1
  Change at Day 1 Cycle 37 |  | -3.00 (NA) — Standard deviation could not be estimated as there was only 1 subject analyzed at the specified time point.
  Change at EOT: number analyzed (Participants) | 28 | 75
  Change at EOT | -8.18 (16.410) | -10.42 (16.256)

9. Secondary Outcome: Number of Subjects With Treatment-Emergent Adverse Events (TEAEs), Serious TEAEs, TEAEs Leading to Discontinuation or TEAEs Leading to Death
Description: AE was defined as any untoward medical occurrence which does not necessarily have a causal relationship with this the study drug. An AE was defined as any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of study drug, whether or not considered related to the study drug. A serious AE was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. Treatment-emergent are events between first dose of study drug and up to 33 days after last dose that were absent before treatment or that worsened relative to pre-treatment state. TEAEs include both Serious TEAEs and non-serious TEAEs. TEAEs were to be reported separately for dacarbazine, pimasertib and pimasertib (crossover) reporting arms.
Time Frame: Baseline up to cut-off date (04-Jul-2015)
Population: Safety analysis set (SAF) consisted of all subjects who received at least 1 dose of any trial treatment.
Measure: Number; unit: subjects
Arm/Group | Dacarbazine | Pimasertib | Pimasertib (Crossover)
Number analyzed (Participants) | 61 | 130 | 41
subjects
  TEAEs | 60 | 130 | 41
  Serious TEAEs | 12 | 74 | 26
  TEAEs Leading to Discontinuation | 3 | 61 | 16
  TEAEs Leading To Death | 4 | 6 | 6

10. Secondary Outcome: Number of Subjects With Adverse Events (AEs) of Special Interest
Description: Adverse events of special interest included ocular retinal vein occlusion, serious retinal detachment or similar retinal abnormality characterized by accumulation of serous fluid in the retina, creatine phosphokinase (CPK) elevation and isoenzyme TEAE of Special Interest (Grade >=2) and acute renal failure (Grade >=2). Subjects were presented under 3 reporting groups: Dacarbazine group: for subjects who received at least 1 dose of dacarbazine; Pimasertib group: for subjects who received at least 1 dose of pimasertib; Pimasertib (Crossover) group: for subjects who were initially randomized and received dacarbazine, but crossed over to pimasertib treatment on progression of their disease.
Time Frame: Baseline up to cut-off date (04-Jul-2015)
Population: Safety analysis set (SAF) consisted of all subjects who received at least 1 dose of any trial treatment.
Measure: Number; unit: subjects
Arm/Group | Dacarbazine | Pimasertib | Pimasertib (Crossover)
Number analyzed (Participants) | 61 | 130 | 41
subjects
  Retinal vein occlusion | 0 | 5 | 2
  Serious retinal detachment | 0 | 76 | 21
  CPK/Isoenzyme TEAE of Special Interest (>=Grade 2) | 0 | 74 | 24
  Acute renal failure (Grade >= 2) | 1 | 9 | 2

11. Secondary Outcome: Number of Subjects With Clinically Significant Change From Baseline in Laboratory Parameter, Vital Signs, Electrocardiogram (ECG) and Ophthalmologic Findings
Description: Subjects were presented under 3 reporting groups: Dacarbazine group: for subjects who received at least 1 dose of dacarbazine; Pimasertib group: for subjects who received at least 1 dose of pimasertib; Pimasertib (Crossover) group: for subjects who were initially randomized and received dacarbazine, but crossed over to pimasertib treatment on progression of their disease.
Time Frame: Baseline up to cut-off date (04-Jul-2015)
Population: Safety analysis set (SAF) consisted of all subjects who received at least 1 dose of any trial treatment.
Measure: Number; unit: subjects
Arm/Group | Dacarbazine | Pimasertib | Pimasertib (Crossover)
Number analyzed (Participants) | 61 | 130 | 41
subjects
  Laboratory Parameter | 0 | 0 | 0
  Vital Signs | 0 | 0 | 0
  ECG | 0 | 0 | 0
  Ophthalmologic Findings | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to cut-off date (04-Jul-2015)
Description: Safety analysis set (SAF) consisted of all subjects who received at least 1 dose of any trial treatment. Subjects were presented under 3 reporting groups: Dacarbazine group: for subjects who received at least 1 dose of dacarbazine; Pimasertib group: for subjects who received at least 1 dose of pimasertib; Pimasertib (Crossover) group: for subjects who were initially randomized and received dacarbazine, but crossed over to pimasertib treatment on progression of their disease.
Arm/Group | Dacarbazine | Pimasertib | Pimasertib (Crossover)
Serious Adverse Events (participants affected / at risk) | 12/61 | 74/130 | 26/41
Other Adverse Events (participants affected / at risk) | 59/61 | 130/130 | 41/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dacarbazine (N=61) | Pimasertib (N=130) | Pimasertib (Crossover) (N=41)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 2
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 2 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 2 | 0
Cardiac failure (Cardiac disorders) | 0 | 3 | 1
Cor pulmonale acute (Cardiac disorders) | 0 | 1 | 0
Left ventricular dysfunction (Cardiac disorders) | 0 | 3 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 1 | 0
Pericarditis (Cardiac disorders) | 1 | 0 | 0
Chorioretinopathy (Eye disorders) | 0 | 1 | 1
Cystoid macular oedema (Eye disorders) | 0 | 0 | 1
Macular detachment (Eye disorders) | 0 | 0 | 1
Macular oedema (Eye disorders) | 0 | 3 | 0
Retinal detachment (Eye disorders) | 0 | 4 | 1
Retinal vein occlusion (Eye disorders) | 0 | 4 | 1
Ulcerative keratitis (Eye disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 6 | 1
Duodenal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 3 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 2
Vomiting (Gastrointestinal disorders) | 1 | 3 | 1
Chest pain (General disorders) | 0 | 1 | 0
Chills (General disorders) | 0 | 1 | 0
Cyst rupture (General disorders) | 0 | 1 | 0
Death (General disorders) | 0 | 1 | 0
Disease progression (General disorders) | 1 | 2 | 1
Fatigue (General disorders) | 0 | 1 | 0
General physical health deterioration (General disorders) | 1 | 2 | 4
Impaired healing (General disorders) | 0 | 1 | 0
Malaise (General disorders) | 0 | 1 | 1
Necrosis (General disorders) | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 4 | 0
Sudden death (General disorders) | 0 | 2 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 1 | 0
Hepatotoxicity (Hepatobiliary disorders) | 0 | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 1 | 0
Candida infection (Infections and infestations) | 0 | 1 | 0
Catheter site infection (Infections and infestations) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 3 | 0
Device related infection (Infections and infestations) | 0 | 1 | 0
Erysipelas (Infections and infestations) | 0 | 7 | 1
Infection (Infections and infestations) | 0 | 1 | 0
Localised infection (Infections and infestations) | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 2 | 1
Septic shock (Infections and infestations) | 0 | 1 | 1
Skin infection (Infections and infestations) | 0 | 1 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 1 | 0
Streptococcal sepsis (Infections and infestations) | 1 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 2 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 26 | 8
Blood creatinine increased (Investigations) | 1 | 0 | 0
Ejection fraction decreased (Investigations) | 0 | 5 | 1
Lipase increased (Investigations) | 0 | 1 | 0
Troponin increased (Investigations) | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Inguinal mass (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Ataxia (Nervous system disorders) | 0 | 1 | 0
Epilepsy (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 0
Metabolic encephalopathy (Nervous system disorders) | 0 | 1 | 0
Neuralgia (Nervous system disorders) | 0 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 1 | 0
Presyncope (Nervous system disorders) | 0 | 2 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 1 | 0
Breast haematoma (Reproductive system and breast disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 5 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 2
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin toxicity (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 1 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 2 | 0
Venous thrombosis limb (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dacarbazine (N=61) | Pimasertib (N=130) | Pimasertib (Crossover) (N=41)
Anaemia (Blood and lymphatic system disorders) | 8 | 13 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 12 | 8 | 3
Neutropenia (Blood and lymphatic system disorders) | 13 | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 1 | 9 | 2
Leukopenia (Blood and lymphatic system disorders) | 6 | 1 | 0
Retinal detachment (Eye disorders) | 0 | 56 | 15
Vision blurred (Eye disorders) | 0 | 29 | 9
Eyelid oedema (Eye disorders) | 1 | 18 | 2
Visual impairment (Eye disorders) | 0 | 12 | 2
Periorbital oedema (Eye disorders) | 0 | 12 | 1
Macular detachment (Eye disorders) | 0 | 10 | 2
Diarrhoea (Gastrointestinal disorders) | 10 | 106 | 31
Nausea (Gastrointestinal disorders) | 25 | 47 | 17
Vomiting (Gastrointestinal disorders) | 14 | 30 | 16
Constipation (Gastrointestinal disorders) | 21 | 24 | 7
Abdominal pain (Gastrointestinal disorders) | 10 | 31 | 7
Dry mouth (Gastrointestinal disorders) | 2 | 20 | 8
Stomatitis (Gastrointestinal disorders) | 3 | 21 | 4
Dyspepsia (Gastrointestinal disorders) | 0 | 11 | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 5 | 2
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 8 | 1
Mouth ulceration (Gastrointestinal disorders) | 0 | 7 | 1
Oedema peripheral (General disorders) | 6 | 59 | 18
Fatigue (General disorders) | 23 | 39 | 11
Asthenia (General disorders) | 13 | 39 | 10
Pyrexia (General disorders) | 5 | 27 | 10
Chills (General disorders) | 3 | 11 | 3
Blood creatine phosphokinase increased (Investigations) | 3 | 86 | 28
Aspartate aminotransferase increased (Investigations) | 3 | 17 | 4
Ejection fraction decreased (Investigations) | 0 | 13 | 3
Weight decreased (Investigations) | 2 | 8 | 3
Alanine aminotransferase increased (Investigations) | 4 | 6 | 1
Weight increased (Investigations) | 0 | 9 | 2
Blood alkaline phosphatase increased (Investigations) | 2 | 5 | 3
Gamma-glutamyltransferase increased (Investigations) | 2 | 4 | 3
Decreased appetite (Metabolism and nutrition disorders) | 8 | 22 | 7
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 13 | 5
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 10 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 4 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 7 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 18 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 9 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 8 | 8
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 9 | 6
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 8 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 3 | 3 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 4
Dizziness (Nervous system disorders) | 3 | 17 | 5
Headache (Nervous system disorders) | 8 | 16 | 0
Dysgeusia (Nervous system disorders) | 6 | 11 | 4
Paraesthesia (Nervous system disorders) | 9 | 4 | 2
Sciatica (Nervous system disorders) | 3 | 5 | 3
Dysaesthesia (Nervous system disorders) | 4 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 5 | 46 | 18
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 47 | 9
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 17 | 7
Erythema (Skin and subcutaneous tissue disorders) | 2 | 14 | 4
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 17 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 13 | 4
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 12 | 6
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 11 | 3
Eczema (Skin and subcutaneous tissue disorders) | 0 | 8 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 4 | 3
Anaemia of chronic disease (Blood and lymphatic system disorders) | 1 | 0 | 0
Eosinophilia (Blood and lymphatic system disorders) | 1 | 0 | 1
Hypochromic anaemia (Blood and lymphatic system disorders) | 0 | 2 | 0
Increased tendency to bruise (Blood and lymphatic system disorders) | 0 | 1 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 2 | 1
Lymph node pain (Blood and lymphatic system disorders) | 1 | 0 | 0
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 2 | 0
Lymphocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 2 | 2 | 1
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 2 | 0
Aortic valve disease (Cardiac disorders) | 0 | 1 | 0
Aortic valve incompetence (Cardiac disorders) | 0 | 3 | 2
Aortic valve stenosis (Cardiac disorders) | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 2 | 0
Atrioventricular block (Cardiac disorders) | 0 | 3 | 0
Atrioventricular block first degree (Cardiac disorders) | 1 | 0 | 1
Atrioventricular block second degree (Cardiac disorders) | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 2 | 1
Bundle branch block (Cardiac disorders) | 0 | 1 | 0
Bundle branch block right (Cardiac disorders) | 0 | 2 | 0
Diastolic dysfunction (Cardiac disorders) | 0 | 1 | 0
Left ventricular dysfunction (Cardiac disorders) | 0 | 4 | 0
Left ventricular hypertrophy (Cardiac disorders) | 0 | 1 | 0
Mitral valve incompetence (Cardiac disorders) | 0 | 4 | 2
Mitral valve sclerosis (Cardiac disorders) | 0 | 0 | 1
Palpitations (Cardiac disorders) | 2 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 1
Pulmonary valve incompetence (Cardiac disorders) | 0 | 1 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 3 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 2
Tachycardia (Cardiac disorders) | 0 | 1 | 0
Tricuspid valve incompetence (Cardiac disorders) | 0 | 5 | 4
Ventricular hypokinesia (Cardiac disorders) | 0 | 0 | 1
Optic nerve hypoplasia (Congenital, familial and genetic disorders) | 0 | 0 | 1
Ventricular septal defect (Congenital, familial and genetic disorders) | 0 | 1 | 0
Cerumen impaction (Ear and labyrinth disorders) | 0 | 1 | 0
Ear congestion (Ear and labyrinth disorders) | 0 | 1 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 3 | 0
Hypoacusis (Ear and labyrinth disorders) | 1 | 0 | 0
Middle ear inflammation (Ear and labyrinth disorders) | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 2 | 1
Vertigo (Ear and labyrinth disorders) | 2 | 3 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 1 | 0
Hyperthyroidism (Endocrine disorders) | 1 | 0 | 0
Blepharitis (Eye disorders) | 0 | 1 | 0
Blindness (Eye disorders) | 0 | 0 | 1
Cataract (Eye disorders) | 0 | 1 | 1
Chalazion (Eye disorders) | 0 | 1 | 0
Chorioretinopathy (Eye disorders) | 0 | 3 | 0
Chromatopsia (Eye disorders) | 0 | 2 | 0
Colour blindness acquired (Eye disorders) | 0 | 1 | 1
Conjunctival haemorrhage (Eye disorders) | 0 | 1 | 0
Conjunctival oedema (Eye disorders) | 0 | 2 | 0
Cystoid macular oedema (Eye disorders) | 0 | 1 | 1
Deposit eye (Eye disorders) | 0 | 1 | 0
Detachment of retinal pigment epithelium (Eye disorders) | 0 | 3 | 2
Diplopia (Eye disorders) | 0 | 1 | 0
Dry eye (Eye disorders) | 1 | 5 | 0
Erythema of eyelid (Eye disorders) | 0 | 1 | 0
Eye discharge (Eye disorders) | 0 | 1 | 0
Eye disorder (Eye disorders) | 0 | 2 | 0
Eye haemorrhage (Eye disorders) | 0 | 1 | 0
Eye inflammation (Eye disorders) | 0 | 1 | 0
Eye oedema (Eye disorders) | 0 | 1 | 0
Eye pain (Eye disorders) | 1 | 3 | 0
Eye pruritus (Eye disorders) | 1 | 0 | 0
Eye swelling (Eye disorders) | 0 | 2 | 0
Eyelid haematoma (Eye disorders) | 0 | 1 | 0
Eyelid ptosis (Eye disorders) | 0 | 3 | 0
Glaucoma (Eye disorders) | 0 | 1 | 0
Lacrimation increased (Eye disorders) | 0 | 3 | 0
Macular cyst (Eye disorders) | 0 | 0 | 1
Macular degeneration (Eye disorders) | 0 | 2 | 0
Macular fibrosis (Eye disorders) | 0 | 4 | 0
Macular oedema (Eye disorders) | 0 | 6 | 1
Myopia (Eye disorders) | 0 | 1 | 0
Ocular hyperaemia (Eye disorders) | 1 | 1 | 0
Ocular hypertension (Eye disorders) | 0 | 3 | 2
Optic disc haemorrhage (Eye disorders) | 0 | 1 | 0
Photophobia (Eye disorders) | 0 | 2 | 0
Photopsia (Eye disorders) | 0 | 2 | 0
Presbyopia (Eye disorders) | 0 | 1 | 0
Retinal deposits (Eye disorders) | 0 | 1 | 0
Retinal disorder (Eye disorders) | 0 | 0 | 2
Retinal haemorrhage (Eye disorders) | 0 | 1 | 0
Retinal oedema (Eye disorders) | 0 | 0 | 1
Retinal pigment epitheliopathy (Eye disorders) | 0 | 2 | 0
Retinal vein occlusion (Eye disorders) | 0 | 1 | 1
Retinopathy (Eye disorders) | 0 | 1 | 0
Subretinal fluid (Eye disorders) | 0 | 1 | 1
Visual acuity reduced (Eye disorders) | 0 | 5 | 0
Vitreous detachment (Eye disorders) | 0 | 1 | 0
Vitreous floaters (Eye disorders) | 0 | 1 | 0
Xerophthalmia (Eye disorders) | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 4 | 2
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 3 | 2
Anal polyp (Gastrointestinal disorders) | 0 | 1 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 4 | 2
Aptyalism (Gastrointestinal disorders) | 0 | 1 | 1
Ascites (Gastrointestinal disorders) | 0 | 2 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 4 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 5 | 2
Epigastric discomfort (Gastrointestinal disorders) | 1 | 0 | 1
Faeces discoloured (Gastrointestinal disorders) | 0 | 2 | 0
Flatulence (Gastrointestinal disorders) | 0 | 2 | 1
Gastric ulcer (Gastrointestinal disorders) | 1 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 2 | 0
Gastritis erosive (Gastrointestinal disorders) | 0 | 1 | 0
Glossitis (Gastrointestinal disorders) | 0 | 2 | 1
Glossodynia (Gastrointestinal disorders) | 0 | 2 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 1 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 2 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 4 | 1
Hyperchlorhydria (Gastrointestinal disorders) | 0 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Lip dry (Gastrointestinal disorders) | 0 | 1 | 0
Lip oedema (Gastrointestinal disorders) | 0 | 1 | 1
Lip pain (Gastrointestinal disorders) | 1 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 1
Mesenteric vein thrombosis (Gastrointestinal disorders) | 0 | 1 | 0
Mouth swelling (Gastrointestinal disorders) | 0 | 0 | 1
Odynophagia (Gastrointestinal disorders) | 0 | 4 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 1 | 0
Oral discomfort (Gastrointestinal disorders) | 0 | 1 | 0
Oral dysaesthesia (Gastrointestinal disorders) | 0 | 1 | 0
Oral mucosal eruption (Gastrointestinal disorders) | 0 | 1 | 0
Oral mucosal erythema (Gastrointestinal disorders) | 0 | 1 | 0
Oral pain (Gastrointestinal disorders) | 0 | 1 | 0
Oral pruritus (Gastrointestinal disorders) | 0 | 1 | 0
Oral toxicity (Gastrointestinal disorders) | 0 | 1 | 0
Paraesthesia oral (Gastrointestinal disorders) | 0 | 1 | 0
Regurgitation (Gastrointestinal disorders) | 1 | 0 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 1 | 0 | 0
Subileus (Gastrointestinal disorders) | 0 | 1 | 0
Tongue disorder (Gastrointestinal disorders) | 0 | 2 | 0
Tongue oedema (Gastrointestinal disorders) | 0 | 0 | 1
Tongue ulceration (Gastrointestinal disorders) | 0 | 2 | 0
Toothache (Gastrointestinal disorders) | 0 | 2 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 1
Axillary pain (General disorders) | 1 | 1 | 1
Catheter site pain (General disorders) | 1 | 0 | 0
Chest discomfort (General disorders) | 1 | 0 | 0
Chest pain (General disorders) | 3 | 2 | 1
Crying (General disorders) | 0 | 1 | 0
Disease progression (General disorders) | 0 | 0 | 1
Drug intolerance (General disorders) | 0 | 1 | 0
Enanthema (General disorders) | 0 | 1 | 0
Face oedema (General disorders) | 0 | 12 | 9
Facial pain (General disorders) | 0 | 0 | 1
Feeling cold (General disorders) | 0 | 3 | 0
Gait disturbance (General disorders) | 0 | 0 | 1
General physical health deterioration (General disorders) | 0 | 2 | 0
Generalised oedema (General disorders) | 0 | 1 | 0
Hyperpyrexia (General disorders) | 0 | 1 | 0
Hyperthermia (General disorders) | 1 | 0 | 0
Hypothermia (General disorders) | 0 | 1 | 1
Inflammation (General disorders) | 0 | 1 | 0
Influenza like illness (General disorders) | 1 | 3 | 0
Injection site haematoma (General disorders) | 0 | 0 | 1
Localised oedema (General disorders) | 0 | 1 | 0
Malaise (General disorders) | 2 | 5 | 2
Mucosal dryness (General disorders) | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 1
Oedema (General disorders) | 0 | 2 | 1
Pain (General disorders) | 0 | 1 | 0
Papillitis (General disorders) | 0 | 1 | 0
Peripheral swelling (General disorders) | 0 | 5 | 2
Secretion discharge (General disorders) | 1 | 0 | 0
Sensation of foreign body (General disorders) | 0 | 1 | 0
Temperature intolerance (General disorders) | 0 | 0 | 1
Vessel puncture site haematoma (General disorders) | 1 | 0 | 0
Vessel puncture site inflammation (General disorders) | 1 | 0 | 0
Vessel puncture site pain (General disorders) | 1 | 0 | 0
Xerosis (General disorders) | 0 | 1 | 2
Cholestasis (Hepatobiliary disorders) | 1 | 4 | 0
Hepatic pain (Hepatobiliary disorders) | 0 | 1 | 0
Hepatocellular injury (Hepatobiliary disorders) | 0 | 7 | 0
Hepatomegaly (Hepatobiliary disorders) | 0 | 1 | 0
Sarcoidosis (Immune system disorders) | 0 | 1 | 0
Abdominal wall abscess (Infections and infestations) | 0 | 0 | 1
Abscess limb (Infections and infestations) | 0 | 0 | 1
Acute sinusitis (Infections and infestations) | 1 | 0 | 0
Acute tonsillitis (Infections and infestations) | 0 | 3 | 1
Bacterial infection (Infections and infestations) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 2 | 2
Cholangitis infective (Infections and infestations) | 0 | 1 | 0
Conjunctivitis (Infections and infestations) | 0 | 8 | 0
Conjunctivitis viral (Infections and infestations) | 0 | 1 | 0
Cystitis (Infections and infestations) | 0 | 2 | 0
Enterobacter infection (Infections and infestations) | 0 | 1 | 0
Erysipelas (Infections and infestations) | 0 | 2 | 0
Folliculitis (Infections and infestations) | 1 | 17 | 7
Fungal oesophagitis (Infections and infestations) | 0 | 1 | 0
Fungal skin infection (Infections and infestations) | 0 | 1 | 0
Furuncle (Infections and infestations) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1 | 1
Helicobacter infection (Infections and infestations) | 0 | 1 | 0
Herpes simplex (Infections and infestations) | 0 | 2 | 0
Herpes virus infection (Infections and infestations) | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 2 | 0
Impetigo (Infections and infestations) | 0 | 2 | 0
Infected bites (Infections and infestations) | 0 | 1 | 0
Infection (Infections and infestations) | 0 | 1 | 0
Influenza (Infections and infestations) | 1 | 2 | 0
Klebsiella infection (Infections and infestations) | 0 | 1 | 0
Laryngitis (Infections and infestations) | 0 | 0 | 1
Localised infection (Infections and infestations) | 0 | 2 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Lung infection (Infections and infestations) | 0 | 1 | 0
Lymph gland infection (Infections and infestations) | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 3 | 8 | 2
Oral candidiasis (Infections and infestations) | 0 | 5 | 1
Oral fungal infection (Infections and infestations) | 0 | 0 | 1
Oral herpes (Infections and infestations) | 0 | 2 | 0
Paronychia (Infections and infestations) | 0 | 9 | 3
Pharyngitis (Infections and infestations) | 0 | 2 | 0
Pneumonia escherichia (Infections and infestations) | 0 | 1 | 0
Pseudomonas infection (Infections and infestations) | 0 | 1 | 1
Pulpitis dental (Infections and infestations) | 0 | 1 | 0
Rash pustular (Infections and infestations) | 1 | 16 | 3
Rhinitis (Infections and infestations) | 1 | 1 | 2
Sinusitis (Infections and infestations) | 1 | 0 | 0
Skin candida (Infections and infestations) | 0 | 2 | 0
Skin infection (Infections and infestations) | 0 | 4 | 1
Staphylococcal bacteraemia (Infections and infestations) | 0 | 1 | 0
Staphylococcal skin infection (Infections and infestations) | 0 | 1 | 0
Superinfection viral (Infections and infestations) | 0 | 1 | 0
Tinea cruris (Infections and infestations) | 0 | 2 | 0
Tinea pedis (Infections and infestations) | 0 | 1 | 0
Tinea versicolour (Infections and infestations) | 0 | 1 | 0
Tonsillitis (Infections and infestations) | 1 | 0 | 0
Tooth abscess (Infections and infestations) | 1 | 0 | 0
Trichophytosis (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 7 | 0
Vaginal infection (Infections and infestations) | 0 | 2 | 0
Viral infection (Infections and infestations) | 1 | 0 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 0 | 1
Wound infection (Infections and infestations) | 1 | 0 | 0
Chest injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 3 | 0
Lip injury (Injury, poisoning and procedural complications) | 0 | 1 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Optic nerve injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 2 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Scratch (Injury, poisoning and procedural complications) | 0 | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Sunburn (Injury, poisoning and procedural complications) | 0 | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Traumatic shock (Injury, poisoning and procedural complications) | 1 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 3 | 0
Wound complication (Injury, poisoning and procedural complications) | 0 | 1 | 0
Amylase increased (Investigations) | 0 | 1 | 1
Blood albumin decreased (Investigations) | 0 | 3 | 0
Blood bicarbonate decreased (Investigations) | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 1 | 1 | 0
Blood creatinine increased (Investigations) | 2 | 2 | 1
Blood fibrinogen decreased (Investigations) | 0 | 1 | 0
Blood lactate dehydrogenase increased (Investigations) | 1 | 3 | 1
Blood phosphorus increased (Investigations) | 0 | 1 | 0
Blood potassium increased (Investigations) | 0 | 1 | 0
Blood pressure increased (Investigations) | 2 | 0 | 0
Blood urea increased (Investigations) | 0 | 1 | 0
Body temperature increased (Investigations) | 1 | 0 | 0
Breath sounds abnormal (Investigations) | 0 | 1 | 0
C-reactive protein increased (Investigations) | 0 | 2 | 0
Creatinine renal clearance decreased (Investigations) | 0 | 1 | 0
Electrocardiogram PR prolongation (Investigations) | 0 | 1 | 0
Electrocardiogram QRS complex prolonged (Investigations) | 0 | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 4 | 1
Electrocardiogram repolarisation abnormality (Investigations) | 0 | 1 | 0
Glomerular filtration rate decreased (Investigations) | 0 | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 2 | 0
Hepatic enzyme increased (Investigations) | 1 | 1 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 1
Intraocular pressure increased (Investigations) | 0 | 3 | 1
Lipase increased (Investigations) | 1 | 2 | 2
Lymphocyte count decreased (Investigations) | 0 | 5 | 0
Neutrophil count decreased (Investigations) | 1 | 3 | 0
Oxygen saturation decreased (Investigations) | 1 | 0 | 0
Platelet count decreased (Investigations) | 1 | 6 | 1
Protein total decreased (Investigations) | 0 | 0 | 1
Protein total increased (Investigations) | 0 | 1 | 0
Pupillary light reflex tests abnormal (Investigations) | 0 | 1 | 0
Troponin increased (Investigations) | 0 | 1 | 0
White blood cell count decreased (Investigations) | 2 | 2 | 0
White blood cell count increased (Investigations) | 0 | 1 | 0
Cell death (Metabolism and nutrition disorders) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 4 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 2 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 1 | 0
Fluid retention (Metabolism and nutrition disorders) | 0 | 2 | 1
Gout (Metabolism and nutrition disorders) | 1 | 1 | 0
Hyperamylasaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 3 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 5 | 0
Hyperlipasaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 3 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 3 | 2
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Increased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0
Iron deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 1 | 1
Oligodipsia (Metabolism and nutrition disorders) | 0 | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Chondrocalcinosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscle contracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Neck mass (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 5 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Trismus (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Blepharal papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 1
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Monoclonal gammopathy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Pyogenic granuloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Ageusia (Nervous system disorders) | 0 | 1 | 0
Altered state of consciousness (Nervous system disorders) | 1 | 0 | 0
Amnesia (Nervous system disorders) | 0 | 2 | 0
Aphasia (Nervous system disorders) | 1 | 1 | 0
Ataxia (Nervous system disorders) | 0 | 1 | 0
Autonomic nervous system imbalance (Nervous system disorders) | 1 | 0 | 0
Balance disorder (Nervous system disorders) | 0 | 1 | 0
Cervicobrachial syndrome (Nervous system disorders) | 0 | 1 | 0
Cognitive disorder (Nervous system disorders) | 0 | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 1 | 0
Dizziness postural (Nervous system disorders) | 0 | 0 | 1
Dysarthria (Nervous system disorders) | 1 | 2 | 0
Hyperaesthesia (Nervous system disorders) | 0 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 1 | 2
Lethargy (Nervous system disorders) | 0 | 2 | 0
Loss of consciousness (Nervous system disorders) | 0 | 2 | 0
Memory impairment (Nervous system disorders) | 0 | 5 | 1
Migraine (Nervous system disorders) | 0 | 0 | 1
Motor dysfunction (Nervous system disorders) | 1 | 0 | 1
Muscle contractions involuntary (Nervous system disorders) | 0 | 1 | 0
Myasthenic syndrome (Nervous system disorders) | 0 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 1 | 1
Neurotoxicity (Nervous system disorders) | 0 | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 2 | 0
Presyncope (Nervous system disorders) | 0 | 3 | 2
Sensorimotor disorder (Nervous system disorders) | 1 | 0 | 0
Sensory disturbance (Nervous system disorders) | 0 | 2 | 1
Somnolence (Nervous system disorders) | 0 | 6 | 1
Syncope (Nervous system disorders) | 0 | 4 | 1
Tremor (Nervous system disorders) | 1 | 2 | 0
Visual field defect (Nervous system disorders) | 0 | 2 | 0
Agitation (Psychiatric disorders) | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 6 | 3 | 2
Confusional state (Psychiatric disorders) | 0 | 3 | 0
Depressed mood (Psychiatric disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 1 | 1 | 0
Dyssomnia (Psychiatric disorders) | 0 | 1 | 0
Euphoric mood (Psychiatric disorders) | 0 | 1 | 0
Hallucination (Psychiatric disorders) | 0 | 1 | 0
Hallucination, visual (Psychiatric disorders) | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 4 | 7 | 1
Irritability (Psychiatric disorders) | 1 | 0 | 0
Mood altered (Psychiatric disorders) | 1 | 0 | 0
Nervousness (Psychiatric disorders) | 0 | 0 | 1
Nightmare (Psychiatric disorders) | 0 | 1 | 0
Persecutory delusion (Psychiatric disorders) | 0 | 1 | 0
Psychomotor retardation (Psychiatric disorders) | 0 | 0 | 2
Acute kidney injury (Renal and urinary disorders) | 0 | 4 | 1
Cystitis noninfective (Renal and urinary disorders) | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 8 | 1
Haematuria (Renal and urinary disorders) | 0 | 2 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 1 | 0
Oliguria (Renal and urinary disorders) | 0 | 2 | 0
Proteinuria (Renal and urinary disorders) | 0 | 4 | 0
Renal injury (Renal and urinary disorders) | 0 | 1 | 0
Renal vein occlusion (Renal and urinary disorders) | 0 | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 2 | 0
Amenorrhoea (Reproductive system and breast disorders) | 0 | 1 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 1 | 0
Genital discomfort (Reproductive system and breast disorders) | 0 | 0 | 1
Genital erythema (Reproductive system and breast disorders) | 1 | 0 | 1
Haematospermia (Reproductive system and breast disorders) | 0 | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 1 | 0
Scrotal haematocoele (Reproductive system and breast disorders) | 0 | 0 | 1
Scrotal oedema (Reproductive system and breast disorders) | 0 | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 9 | 3
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 5 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 26 | 6
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 8 | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nasal disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Nasal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Nocturnal dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 3
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pharyngeal ulceration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 2
Rales (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 3 | 1
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 0 | 2 | 2
Diffuse alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Erythrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hair growth abnormal (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hirsutism (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 2 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 2 | 1
Intertrigo (Skin and subcutaneous tissue disorders) | 1 | 4 | 0
Nail bed inflammation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Onycholysis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 4 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 6 | 0
Papule (Skin and subcutaneous tissue disorders) | 0 | 3 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 2 | 3 | 0
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Prurigo (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 4 | 2
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 5 | 1
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 2 | 1
Rash morbilliform (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 4 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rosacea (Skin and subcutaneous tissue disorders) | 1 | 2 | 1
Scab (Skin and subcutaneous tissue disorders) | 1 | 2 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin burning sensation (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Skin erosion (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 4 | 1
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin mass (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Solar dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 4 | 0
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Capillary leak syndrome (Vascular disorders) | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0
Diastolic hypertension (Vascular disorders) | 0 | 1 | 0
Flushing (Vascular disorders) | 2 | 1 | 1
Haematoma (Vascular disorders) | 2 | 1 | 0
Hot flush (Vascular disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 2 | 21 | 6
Hypotension (Vascular disorders) | 3 | 4 | 2
Lymphoedema (Vascular disorders) | 2 | 11 | 3
Pelvic venous thrombosis (Vascular disorders) | 0 | 1 | 0
Peripheral coldness (Vascular disorders) | 0 | 1 | 0
Peripheral ischaemia (Vascular disorders) | 0 | 0 | 1
Peripheral venous disease (Vascular disorders) | 1 | 0 | 0
Phlebitis (Vascular disorders) | 0 | 0 | 1
Thrombophlebitis (Vascular disorders) | 0 | 1 | 0
Vascular compression (Vascular disorders) | 1 | 0 | 0
Vena cava thrombosis (Vascular disorders) | 1 | 0 | 0
Venous thrombosis limb (Vascular disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other